CLINICAL TRIAL: NCT00103987
Title: Neurobiological Mechanisms in Panic Disorder: Behavioral, Genetic, & Neural Correlates of Noradrenergic Function
Brief Title: Neurobiological Mechanisms in Panic Disorder
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050102; 05-M-0102
Record Dates: First submitted 2005-02-17; First posted 2005-02-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-11-12

CONDITIONS: Panic Disorder
Keywords: Panic Disorder; Norepinephrine; Yohimbine; Genes; Pathophysiology; Noradrenergic Mechanisms; PET Imaging; PD; Healthy Volunteer; HV
MeSH Terms: conditions — Panic Disorder

SUMMARY:
This study will examine brain and noradrenaline function in panic disorder. Noradrenaline is a brain chemical that is involved in the regulation of emotion, anxiety, sleep, stress hormones such as cortisol, and other body functions that are disturbed in panic disorder.

Healthy normal volunteers and patients with panic disorder between 18 and 60 years of age may be eligible for this study. Candidates are screened with psychiatric and medical histories, a physical examination, blood and urine tests, and an electrocardiogram.

Participants undergo the following tests and procedures:

* Blood draw to obtain DNA for genetic studies of panic disorder - particularly of a gene that helps control noradrenaline activity - and to grow cell lines that can be frozen and used for future research on the disorder.
* Magnetic resonance imaging: MRI uses a magnetic field and radio waves to produce images of body tissues and organs. For this procedure, the subject lies on a table that is moved into the scanner (a narrow cylinder), and wears earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. The procedure lasts about 60 minutes, during which the patient is asked to lie still for 10 to 15 minutes at a time.
* Yohimbine injection with PET scanning: Catheters (plastic tubes) are placed in two veins, one to administer yohimbine, a drug that increases noradrenaline activity in the body for about 60 minutes, and one to draw blood samples. Yohimbine often causes temporary trembling, goosebumps, and clammy palms, and may cause emotions such as elation, anxiety, panic attacks, or depression. During yohimbine administration, subjects undergo positron emission tomography (PET) scanning. PET uses small amounts of a radioactive chemical called [fluoro-18]-fluorodeoxyglucose that "labels" active areas of the brain, showing patterns of glucose (sugar) metabolism. For the procedure, the subject lies on the scanner bed, with a special mask fitted to his or her head and attached to the bed to help keep the head still. A brief "transmission" scan is done just before the radioactive tracer is injected in order to calibrate the scanner. After the tracer is injected through the catheter, pictures are taken for about an hour, while the subject lies still on the scanner bed.
* Saline injection with PET scanning: The procedure is the same as that described above, except a saline solution is administered as placebo instead of yohimbine.

DETAILED DESCRIPTION:
A considerable body of preclinical and clinical evidence suggests that dysregulated activity of noradrenergic systems in the brain is involved in the development of mood disturbance, anxiety, and fear. Neuroanatomical and neurophysiological studies of the noradrenergic system provide a basis for relating increased activity of this system to the behavioral expression of fear and anxiety and the somatic symptoms and cardiovascular changes that accompany severe anxiety states. Previously, extensive research has been done on the role of noradrenergic mechanisms in panic disorder (PD), and it has been suggested that in at least a subgroup of PD patients an abnormality of noradrenergic mechanisms may exist. Studies in patients with PD using the alpha2-adrenoreceptor (AR) antagonist yohimbine showed that a subgroup of PD patients exhibit abnormalities in the regulation of noradrenergic function. Yohimbine, which activates noradrenergic neurons, has been shown to produce greater increases in anxiety, somatic symptoms, blood pressure and plasma levels of the noradrenergic metabolite MHPG in some patients with PD relative to healthy controls. The effect of yohimbine on brain regions hypothesized to be involved in the pathogenesis of PD has not been determined in PD patients using modern neuroimaging techniques. The anxiogenic effects of yohimbine do not occur in all PD patients, although the neurobiological basis for this differential response to yohimbine has not been identified.

This research project proposes to address these two unresolved questions. The effects of yohimbine on regional cerebral glucose metabolism will be determined in PD patients and healthy controls. In addition, preliminary data will be obtained as to whether the behavioral and cerebral metabolic responses to yohimbine relate to functional polymorphisms of the COMT gene which affect catecholamine metabolism.

It is predicted that yohimbine will produce decreases in cerebral metabolism in the prefrontal cortex, orbitofrontal cortex, and anterior cingulate. Healthy controls will exhibit an inverse direction of change in these brain regions. These findings would be similar to those we have previously observed in PTSD patients and may reflect an altered dose-response effect of yohimbine in PD and PTSD relative to controls since preclinical pharmacological studies of stress have shown that high levels of norepinephrine release in the brain decrease brain metabolism whereas lower levels increase brain metabolism. In terms of polymorphisms of the COMT and other catecholamine systems-related gene polymorphisms, it is predicted that the low-activity COMT (met allele) alleles will be associated with greater behavioral and cerebral metabolic responses to yohimbine.

ELIGIBILITY:
* INCLUSION CRITERIA:

Up to 120 drug-free subjects (ages 18-60) will be selected who additionally meet criteria for one of 3 subgroups:

I. PD, current (n=30), as defined by DSM-IV criteria for PD, and still symptomatic as defined by at least 1 panic attack/week or a CGI score of at least 4. In case of co-morbid depression it will be ensured that PD is the primary diagnosis. This means that PD preceded the onset of MDD. These patients will be drug-free for at least 2 weeks prior to being enrolled in the study.

II. PD, remitted (n=30), as defined by DSM-IV criteria for PD, and asymptomatic as no longer meeting criteria for PD while being drug-free during the past 6 months.

III. Healthy Control Sample. Sixty subjects (ages 18-60) who have not met criteria for any major psychiatric disorder (axis I diagnosis according to DSM-IV). A control subject will be matched to each PD subject for age, gender, menopausal and estrogen replacement status, and handedness. The control subjects will have no known first-degree relatives with any axis I disorder.

EXCLUSION CRITERIA:

Symptomatic PD patients must not have taken any antidepressant or other medications likely to alter monoamine neurochemistry or cerebrovascular and cardiovascular function for at least 2 weeks prior to the challenge studies.

Remitted PD patients will be drug-free for at least 6 months prior to enrollment.

Subjects will also be excluded if they have:

1. evidence for an axis I psychiatric disorder (DSM-IV criteria) other than panic disorder with/without agoraphobia with/without comorbid depression,
2. medical or neurological illnesses likely to affect physiology or anatomy, i.e. hypertension, cardiovascular disorders, seizures,
3. a history of drug (including BZDs) or alcohol abuse within 1 year or a lifetime history of alcohol or drug dependence (DSM IV criteria),
4. current pregnancy (as documented by pregnancy testing at screening or on the days of the challenge studies),
5. current breast feeding,
6. are smokers,
7. presence of an axis II personality disorder,
8. current treatment with fluoxetine, or
9. history of an adverse reaction associated with the administration of yohimbine.

Subjects beyond age 60 are excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2005-02-14; Study Completion 2010-11-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bisaga A, Katz JL, Antonini A, Wright CE, Margouleff C, Gorman JM, Eidelberg D. Cerebral glucose metabolism in women with panic disorder. Am J Psychiatry. 1998 Sep;155(9):1178-83. doi: 10.1176/ajp.155.9.1178. PMID 9734539
- [Background] Cameron OG, Zubieta JK, Grunhaus L, Minoshima S. Effects of yohimbine on cerebral blood flow, symptoms, and physiological functions in humans. Psychosom Med. 2000 Jul-Aug;62(4):549-59. doi: 10.1097/00006842-200007000-00014. PMID 10949101
- [Background] Schmidt ME, Oshinsky RJ, Kim HG, Schouten JL, Folley BS, Potter WZ. Cerebral glucose metabolic and plasma catecholamine responses to the alpha(2) adrenoceptor antagonist ethoxyidazoxan given to healthy volunteers. Psychopharmacology (Berl). 1999 Sep;146(2):119-27. doi: 10.1007/s002130051097. PMID 10525746